CLINICAL TRIAL: NCT00652496
Title: Safety and Efficacy Study of Different Formulations of Bimatoprost Once-Daily in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-030
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental): Bimatoprost 0.01% ophthalmic solution
  Interventions: Drug: Bimatoprost 0.01% ophthalmic solution
- 2 (Experimental): Bimatoprost 0.015% formulation 1 ophthalmic solution
  Interventions: Drug: Bimatoprost 0.015% formulation 1 ophthalmic solution
- 3 (Experimental): Bimatoprost 0.015% formulation 2 ophthalmic solution
  Interventions: Drug: Bimatoprost 0.015% formulation 2 ophthalmic solution
- 4 (Experimental): Bimatoprost 0.02% ophthalmic solution
  Interventions: Drug: Bimatoprost 0.02% ophthalmic solution
- 5 (Active Comparator): Bimatoprost 0.03% ophthalmic solution
  Interventions: Drug: Bimatoprost 0.03% ophthalmic solution

INTERVENTIONS:
Drug: Bimatoprost 0.01% ophthalmic solution — One drop in one eye, once daily in the morning for 4 consecutive days, the other eye received the active control eye drop
  Arms: 1
Drug: Bimatoprost 0.015% formulation 1 ophthalmic solution — One drop in one eye, once daily in the morning for 4 consecutive days, the other eye received the active control eye drop
  Arms: 2
Drug: Bimatoprost 0.015% formulation 2 ophthalmic solution — One drop in one eye, once daily in the morning for 4 consecutive days, the other eye received the active control eye drop
  Arms: 3
Drug: Bimatoprost 0.02% ophthalmic solution — One drop in one eye, once daily in the morning for 4 consecutive days, the other eye received the active control eye drop
  Arms: 4
Drug: Bimatoprost 0.03% ophthalmic solution — Bimatoprost 0.03% ophthalmic solution, one drop in one eye, once daily in the morning for 4 consecutive days, the other eye received one drop of any of the 4 study drugs
  Other Names: LUMIGAN®
  Arms: 5

SUMMARY:
This study evaluates the safety and efficacy of different formulations of bimatoprost ophthalmic solution compared with Bimatoprost 0.03% once-daily in patients with glaucoma or ocular hypertension. One of the test formulations was given to one eye and bimatoprost 0.03% given to the fellow eye of each patient

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or glaucoma in both eyes
* Require IOP-lowering therapy in each eye

Exclusion Criteria:

* Uncontrolled systemic disease
* Known allergy or hypersensitivity to bimatoprost

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2005-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | Day 5

SECONDARY OUTCOMES:
Patient Comfort | Days 1-4
Patient Satisfaction | Day 5
Treatment Preference | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Wenatchee, Washington, United States